CLINICAL TRIAL: NCT05108558
Title: Efficacy of a Novel Collagenase Clostridium Histolyticum Protocol for Peyronie's Disease Among Prior Non-responders: A Randomized, Controlled, Single-Blinded Study
Brief Title: Efficacy of a Novel CCH Protocol for PD Among Prior Non-responders
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Charitable Union for the Research and Education of Peyronie's Disease (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUREPD 103
Record Dates: First submitted 2021-10-11; First posted 2021-11-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Peyronie's Disease
MeSH Terms: conditions — Penile Induration | interventions — Microbial Collagenase

STUDY DESIGN:
Intervention Model Description: Patients meeting criteria who have consented will be randomized to either control or CCH x 6 months, followed by a cross-over phase where controls will receive CCH. See Figure 1 for full study schema.
  1. Control. Men in this cohort would undergo baseline assessments followed by no treatment for 6 months and then repeat assessments. Men would then cross-over to the CCH treatment phase and undergo up to 8 injections (or until curvature is <15 degrees, whichever comes first). Final assessments would then be performed 6 weeks following the final injection.
  2. CCH followed by observation. Men in this cohort would undergo baseline assessments followed by up to 8 injections of CCH (or until curvature is <15 degrees). Assessments would then be performed 6 weeks after completion of treatment. Men then would not undergo any additional treatments for 6 months, after which they would have final assessments performed.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Photography will be obtained where possible, with outcomes assessed based on the photographs. The care provider obtaining measurements will also be blinded as to baseline outcomes and results with follow-up assessments.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control - Crossover to CCH (Active Comparator): Men in this cohort would undergo baseline assessments followed by no treatment for 6 months and then repeat assessments. Men would then cross-over to CCH treatment and undergo up to 8 injections (or until curvature is <15 degrees). Final assessments would then be performed 6 weeks following the final injection.
  Interventions: Drug: Control - Crossover to CCH; Device: RestoreX
- Collagenase Clostridium Histolyticum (Experimental): Men in this cohort would undergo baseline assessments followed by up to 8 injections of CCH (or until curvature is <15 degrees). Men would then undergo assessments 6 weeks later, followed by a 6-month no treatment phase and then final assessments.
  Interventions: Drug: CCH administration; Device: RestoreX

INTERVENTIONS:
Drug: CCH administration — Patients will be randomized 3:1 into the CCH administration arm. After undergoing baseline assessments, this arm will receive up to 8 CCH injections, followed by final assessments 6 weeks later.
  Other Names: Collagenase Clostridium Histolyticum
  Arms: Collagenase Clostridium Histolyticum
Drug: Control - Crossover to CCH — Patients will be randomized 1:3 into the control arm. After undergoing baseline assessments, control men will not undergo treatments for 6 months. They will then have repeat assessments and receive up to 8 CCH injections. They will then have final assessments performed 6 weeks after treatment.
  Other Names: Collagenase Clostridium Histolyticum
  Arms: Control - Crossover to CCH
Device: RestoreX — Both treatment arms will incorporate the use of RestoreX for 30-60 minutes daily during CCH administration and continued until 6 weeks after final injection administration.

SUMMARY:
Compare key clinical outcomes between controls and men treated with a novel CCH administration protocol among men previously unresponsive to CCH administration.

DETAILED DESCRIPTION:
Beginning approximately 3 years ago, the investigators' team sought to achieve further improvements with CCH through the addition of more aggressive modeling therapies. Results from a comparison of CCH alone vs CCH and traction with RestoreX demonstrated a mean 33.8 degree (49%) curvature improvement with combined therapy compared to 19-20 degrees (30-31%) with CCH alone or CCH and other traction devices). These results currently represent the greatest improvements with CCH in published literature and further build upon phase IIb results which demonstrated that mechanical traction (via manual modeling in the phase IIb trial) represents a critical factor in achieving improvements with CCH.

The investigators' team additionally published a survey of men who had experienced suspected penile fractures with CCH and demonstrated greater curvature improvements without any loss / worsening of erectile function. This critical study highlighted that conservative management of suspected fractures should not only be considered a standard of care in managing suspected fractures, but also that these men achieved better final outcomes (again highlighting the importance of the combination of mechanical curvature correction in addition to CCH management).

Based on the above findings, the investigators' team began performing a more aggressive manual modeling protocol. This novel protocol included several notable innovations: dilution of the 0.9 mg of CCH in 0.7 ml of diluent, injection to the erect penis to assure accurate injection, repeat curvature assessments with each series (due to changing of the point of maximal curvature), incorporation of RestoreX traction therapy post injection, and 'aggressive' manual modeling (equivalent of 10-15 lbs of force) to achieve curvature correction. Preliminary (unpublished - abstract submitted to SMSNA 2021) results from these men demonstrated a median ~60% curvature improvement. Importantly, several of the patients had previously undergone 8 CCH injections with outside providers and were able to similarly achieve a median 60% improvement with the investigators' injection / modeling protocol.

These preliminary findings have several important ramifications for the treatment of PD:

1. Men who have previously not achieved adequate curvature correction with 4 series of CCH injections may benefit from additional injections using a more aggressive traction protocol.
2. A more aggressive traction protocol would benefit patients to achieve greater outcomes than with previously reported protocols.

1.2 Investigational Treatments

The current study would randomize men 1:3 into one of two treatment cohorts: 1. Observation followed by CCH or 2. CCH followed by observation. This study design offers the benefits of a randomized, controlled trial (highest level of evidence). RCTs are particularly important in PD, where the disease changes over time in a percentage of men as a function of its natural history. This would also allow blinding of measurements using photographs (single-blinded assessments), which provides further study rigor.

1. No treatment (control) followed by CCH. Men in this cohort would undergo baseline assessments followed by no treatment for 6 months and then repeat assessments. Men would then cross-over to CCH treatment and undergo up to 8 injections (or until curvature is <15 degrees). Interval assessments would be performed with the 1st injection of each series, and final assessments would then be performed 6 weeks following the final injection.
2. CCH followed by no treatment. Men in this cohort would undergo baseline assessments followed by up to 8 injections of CCH (or until curvature is <15 degrees). Interval assessments would be performed with the 1st injection of each series and 6 weeks following completion of treatment. Men then would not undergo any additional treatments for 6 months, after which final assessments would then performed.

ELIGIBILITY:
Inclusion Criteria:

* Men with Peyronie's Disease
* >18 years old
* Curvature ≥30 degrees
* Previously completed 6-8 CCH injections
* Prior minimal (<20% and/or <10 degrees) responsiveness to CCH administration
* Prior CCH injections must have been performed without use of a Restorex traction device and used the IMPRESS protocol
* Ability to achieve an erection satisfactory for intercourse with or without PDE5 inhibitors
* The patient exhibits a palpable plaque consistent with Peyronie's Disease

Exclusion Criteria:

* Prior surgical treatment on the penis (other than circumcision)
* Any contraindications to CCH - as determined by the PI
* Inability to complete 8 additional CCH injections
* Severe plaque calcification (i.e. >1 cm shadowing)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Penile Curvature | 6 months
  Compare the change in degree of penile curvature from baseline (using a goniometer) between control and treatment groups at 6 months
Peyronie's Disease Questionnaire Outcomes | 6 months
  Compare Peyronie's Disease Questionnaire outcomes between control and treatment groups at 6 months using the Peyronie's Disease Questionnaire (15 items; subdomains - psychological and physical (Q1-6, 0-24), penile pain (Q7-9; 0-30), symptom bother (Q10-15; 0-16); 12 and 14 (Y/N q's); lower is better.

SECONDARY OUTCOMES:
International Index of Erectile Function Outcomes | 6 months
  Compare International Index of Erectile Function Outcomes between control and treatment groups at 6 months
Penile Curvature Compared to Baseline | 12 months
  Compare penile curvature changes (degrees) in control men at baseline and 12 months (i.e. prior to and following cross-over to CCH) - using goniometer
Penile Length Compared to Baseline | 12 months
  Compare penile length changes in control men at baseline and 12 months (i.e. prior to and following cross-over to CCH)
Compare Peyronie's Disease Questionnaire to Baseline | 12 months
  Compare PDQ changes in control men at baseline and 12 months (i.e. prior to and following cross-over to CCH) using the Peyronie's Disease Questionnaire (15 items; subdomains - psychological and physical (Q1-6, 0-24), penile pain (Q7-9; 0-30), symptom bother (Q10-15; 0-16); 12 and 14 (Y/N q's); lower is better.
Compare International Index of Erectile Function to baseline | 12 months
  Compare International Index of Erectile Function changes in control men at baseline and 12 months (i.e. prior to and following cross-over to CCH)
Penile Length Between Groups | 6 months
  Compare penile length changes between control and treatment groups at 6 months
Adverse events - 6 months - pain, sensation, swelling | 6 months
  Report adverse events at the 6-month time point
Adverse events - 12 months - pain, sensation, swelling | 12 months
  Report adverse events at the 12-month time point
Change in penile curvature durability | 6 months
  Report changes in penile curvature degree between the 6 and 12-month assessments for CCH men by goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Landon Trost, MD, Principal Investigator — CURE PD
Locations (1):
- The Male Fertility and Peyronie's Clinic, Orem, Utah, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT05108558/Prot_SAP_000.pdf